CLINICAL TRIAL: NCT00175097
Title: Impact of Different Forms of Soybean Based Foods on Cardiovascular Disease Risk Factors in Hypercholesterolemic Subjects.
Brief Title: Soybean Based Diets and CVD Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HL 58008-1785; R01HL058008 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Hypercholesterolemia
Keywords: soy protein; lipids; lipoproteins; apolipoproteins; cholesterol; endothelial function
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- soybeans and products made thereof (Other): Diet: soybeans and products made thereof (soynuts, soynut butter, soy flakes & grits)
  Interventions: Other: Diet: soybeans and products made thereof
- soybean flour and products made thereof (Other): Diet: soybean flour and products made thereof (textured soybean)
  Interventions: Other: Diet: soybean flour and products made thereof
- soybean milk (Other): Diet: soybean milk (tofu, soybean yogurt, cheese, etc.)
  Interventions: Other: Diet: soybean milk
- animal protein based diet (Other): Diet: animal protein based diet
  Interventions: Other: Diet: Animal protein based diet

INTERVENTIONS:
Other: Diet: soybeans and products made thereof — The macronutrient composition of each diets will be similar. The difference will be the type of protein (animal or soybean) or form of soybean incorporated into various food mixtures. This diet will incorporate soybeans and products made thereof.
  Arms: soybeans and products made thereof
Other: Diet: soybean flour and products made thereof — The macronutrient composition of each diets will be similar. The difference will be the type of protein (animal or soybean) or form of soybean incorporated into various food mixtures. This diet will incorporate soybean flour and products made thereof.
  Arms: soybean flour and products made thereof
Other: Diet: soybean milk — The macronutrient composition of each diets will be similar. The difference will be the type of protein (animal or soybean) or form of soybean incorporated into various food mixtures. This diet will incorporate soybean milk.
  Arms: soybean milk
Other: Diet: Animal protein based diet — The macronutrient composition of each diets will be similar. The difference will be the type of protein (animal or soybean) or form of soybean incorporated into various food mixtures. This diet will incorporate animal protein.
  Arms: animal protein based diet

SUMMARY:
To evaluate the impact of soybean processing as well as the effect of soy relative to animal protein, independent of alterations in the fatty acid profile of the diet on CVD risk factors in hypercholesterolemic subjects.

DETAILED DESCRIPTION:
Recent data suggests that the magnitude of the effect of soy protein on lipid and lipoprotein levels is variable and less dramatic than originally reported. This discordance might be attributable to the forms of soy protein used, as well as subtle unrecognized shifts in the fatty acid, cholesterol and fiber content of the diets.The aim of the present investigation is to assess the effects of different forms of soybeans (whole bean and products made thereof), products derived from soy flour (textured soy protein) and products made from a soybean extract (i.e. tofu, yogurt) relative to animal protein, independent of alterations in the fatty acid profile of the diet on CVD risk factors in hypercholesterolemic subjects. The intent is to isolate any potential impact of processing on the plasma lipid lowering efficacy of the soy product or soy protein relative to animal protein.

ELIGIBILITY:
Inclusion Criteria:

Plasma LDL-C >120mg/dL, Free from chronic illness, Not taking medications known to affect lipid metabolism (lipid lowering drugs, beta-blockers, fish-oil capsules, cis-retinoic acid, ascorbic acid, vitamin E, diuretics or hormones), Post-menopausal women.

Exclusion Criteria:

Soy allergy, Smokers, Consuming >2 alcoholic drinks per day, Pre-menopausal women.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2001-06; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Fasting and non-fasting plasma lipids, apolipoproteins; end of each dietary phase | 24 weeks
Vascular endothelial function; end of each dietary phase | 24 weeks
Susceptibility of LDL to oxidation; end of each dietary phase | 24 weeks
C-reactive protein; end of each dietary phase | 24 weeks

SECONDARY OUTCOMES:
Endogenous cholesterol synthesis; end of each dietary phase | 24 weeks
Endogenous triglyceride synthesis; end of each dietary phase | 24 weeks
Plasma and Urinary Isoflavone levels; end of each dietary phase | 24 weeks
Genotyping of candidate genes involved in the variability observed in response to dietary modification | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alice H Lichtenstein, DSc, Principal Investigator — Tufts University (HNRCA)
Locations (2):
- United States (2):
  - Division of Cardiology, Tufts-New England Medical Center Hospitals, Tufts University School of Medicine, Boston, Massachusetts
  - Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts